CLINICAL TRIAL: NCT02123654
Title: A Japanese Phase 3 Study of a Daclatasvir/Asunaprevir/BMS-791325 Fixed Dose Combination (FDC) in Treatment-Naive and IFN Experienced Subjects With Genotype 1 Chronic Hepatitis C
Brief Title: UNITY 3: A Japanese Phase 3 Study of a Daclatasvir/Asunaprevir/BMS-791325 in Subjects With Genotype 1 Chronic Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AI443-117
Record Dates: First submitted 2014-04-10; First posted 2014-04-25 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-08

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; asunaprevir; 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: DCV 3DAA + Placebo for DCV/Placebo for ASV (Experimental): DCV 3DAA tablet orally twice daily for 12 weeks + Placebo for DCV tablet orally once daily and Placebo for ASV capsule orally twice daily for 24 weeks (Double blind)
  Interventions: Drug: DCV 3DAA; Other: Placebo for Daclatasvir; Other: Placebo for Asunaprevir
- Arm 2: DCV/ASV + Placebo for DCV 3DAA (Active Comparator): Daclatasvir 60 mg tablet orally once daily and Asunaprevir 100 mg capsule orally twice daily for 24 weeks + Placebo for DCV 3DAA tablet orally twice daily for 12 weeks (Double blind)
  Interventions: Drug: Daclatasvir; Drug: Asunaprevir; Other: Placebo for DCV 3DAA
- DCV 3DAA (Experimental): DCV 3DAA (open label) Tablet orally twice daily for 12 weeks
  Interventions: Drug: DCV 3DAA

INTERVENTIONS:
Drug: Daclatasvir
  Arms: Arm 2: DCV/ASV + Placebo for DCV 3DAA
Drug: Asunaprevir
  Arms: Arm 2: DCV/ASV + Placebo for DCV 3DAA
Drug: DCV 3DAA
  Other Names: Daclatasvir 30 mg /Asunaprevir 200 mg /BMS-791325 75 mg fixed dose combination
  Arms: Arm 1: DCV 3DAA + Placebo for DCV/Placebo for ASV; DCV 3DAA
Other: Placebo for DCV 3DAA
  Arms: Arm 2: DCV/ASV + Placebo for DCV 3DAA
Other: Placebo for Daclatasvir
  Arms: Arm 1: DCV 3DAA + Placebo for DCV/Placebo for ASV
Other: Placebo for Asunaprevir
  Arms: Arm 1: DCV 3DAA + Placebo for DCV/Placebo for ASV

SUMMARY:
The purpose of this study is to demonstrate that the proportion of treatment-naive non-cirrhotic subjects with Genotype (GT)-1b treated with Daclatasvir (DCV)/Asunaprevir (ASV)/BMS-791325 who achieve Sustained Virologic response (SVR12), defined as Hepatitis C virus (HCV) RNA < LOQ target detected or target not detected (LOQ TD/TND) at follow-up Week 12, is significantly higher than SVR12 of current Standard of Care (SOC).

DETAILED DESCRIPTION:
Limit of Quantitation (LOQ)

Ribonucleic acid (RNA)

End of Treatment (EOT)

Triple Direct Acting Antivirals (3DAA)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Males and females, ≥ 20 years of age
* Subjects chronically infected with HCV GT-1
* HCV RNA viral load of ≥ 100,000 IU/mL

Exclusion Criteria:

* Hepatocellular carcinoma
* Co-infection with Hepatitis B virus (HBV) or Human immunodeficiency virus (HIV)
* Severe or uncontrollable complication

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Proportion of treated subjects who achieve SVR12 in treatment-naive non-cirrhotic subjects treated with DCV/ASV/BMS-791325, defined as HCV RNA < LOQ target detected or target not detected (LOQ TD/TND) at post-treatment follow-up Week 12 | After 12 weeks of the last dose

SECONDARY OUTCOMES:
The proportion of treatment-naive subjects who achieve SVR12 with DCV/ASV/BMS-791325 or DCV/ASV | Weeks: 1, 2, 4, 6, 8, 12, 16, 20 and 24; EOT (week 12 or 24); post-treatment Weeks 4, 8, 12 and 24
The proportion of Interferon (IFN) experienced subjects who achieve SVR12 with DCV/ASV/BMS-791325 | Weeks: 1, 2, 4, 6, 8, 12, 16, 20 and 24; EOT (week 12 or 24); post-treatment Weeks 4, 8, 12 and 24
The proportion of subjects who achieve HCV RNA < LOQ TD/TND at each of the following Weeks: 1, 2, 4, 6, 8, 12, 16, 20 and 24; EOT; post-treatment Weeks 4 (SVR4), 8 (SVR8) and 24 (SVR24) | Weeks: 1, 2, 4, 6, 8, 12, 16, 20 and 24; EOT (week 12 or 24); post-treatment Weeks 4, 8, 12 and 24
The proportion of subjects who achieve HCV RNA < LOQ TND at each of the following Weeks: 1, 2, 4, 6, 8, 12, 16, 20 and 24; EOT; post-treatment Weeks 4, 8, 12 and 24 | Weeks: 1, 2, 4, 6, 8, 12, 16, 20 and 24; EOT (week 12 or 24); post-treatment Weeks 4, 8, 12 and 24
On-treatment safety as measured by the frequency of Serious Adverse Event (SAEs), discontinuations due to Adverse Event (AEs), and selected Grade 3 - 4 laboratory abnormalities | Approximately 48 weeks
  based on the US National Institutes of Health Division of AIDs (DAIDS) criteria
The proportion of subjects with anemia defined as Hb < 10 g/dL on-treatment who had Hb ≥ 10 g/dL at baseline | Approximately 48 weeks
The proportion of subjects in each cohort who achieve SVR12 associated with HCV genotype subtype 1a vs 1b | Weeks: 1, 2, 4, 6, 8, 12, 16, 20 and 24; EOT (week 12 or 24); post-treatment Weeks 4, 8, 12 and 24
The proportion of subjects in each cohort who achieve SVR12 associated with IL28B Single Nucleotide Polymorphisms (SNP) status | Weeks: 1, 2, 4, 6, 8, 12, 16, 20 and 24; EOT (week 12 or 24); post-treatment Weeks 4, 8, 12 and 24
The proportion of cirrhotic and non-cirrhotic subjects who achieve SVR12 | Weeks: 1, 2, 4, 6, 8, 12, 16, 20 and 24; EOT (week 12 or 24); post-treatment Weeks 4, 8, 12 and 24
On-treatment safety of non-cirrhotic vs cirrhotic subjects, as measured by the frequency of SAEs, discontinuations due to AEs, and selected Grade 3 - 4 laboratory abnormalities on DAIDS criteria | Approximately 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (32):
- Japan (32):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Fukui-shi, Fukui
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kurume-shi, Fukuoka
  - Local Institution, Gifu, Gifu
  - Local Institution, Ogaki-shi, Gifu
  - Local Institution, Takasaki, Gunma
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kobe, Hyōgo
  - Local Institution, Kanazawa, Ishikawa-ken
  - Local Institution, Takamatsu, Kagawa-ken
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Kawasaki-shi, Kanagawa
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Kumamoto, Kumamoto
  - Local Institution, Kyoto, Kyoto
  - Local Institution, Miyazaki, Miyazaki
  - Local Institution, Kashihara, Nara
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Osaka, Osaka
  - Local Institution, Suita, Osaka
  - Local Institution, Suita-shi, Osaka
  - Local Institution, Saga, Saga-ken
  - Local Institution, Iruma-gun, Saitama
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Minato-ku, Tokyo
  - Local Institution, Musashino-shi, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo
  - Local Institution, Yamagata, Yamagata
  - Local Institution, Chuo-shi, Yamanashi
  - Local Institution, Nishinomiya-shi

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx